CLINICAL TRIAL: NCT06566144
Title: Effect of a Standard Treatment for Non-specific Low Back Pain Combined With Multimodal Osteopathy Treatment on Pain Intensity and Functional Capacity: A Randomized, Controlled, Blinded Trial"
Brief Title: Standard Treatment for Non-specific Low Back Pain Combined With Multimodal Osteopathy Treatment on Pain Intensity and Functional Capacity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Fabiano Politti, Prof. Fabiano Politti, FT, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FP004
Record Dates: First submitted 2024-08-09; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathy treatment (Experimental): The osteopathy treatment group (OTG) will be submitted to a clinical method considered the gold standard for the treatment of non-specific low back pain together with osteopathy treatment
  Interventions: Other: Osteopathy treatment
- Standard treatment (Active Comparator): The Standard treatment group (STG) will only receive the gold standard method for the treatment of low back pain.
  Interventions: Other: Standard treatment

INTERVENTIONS:
Other: Standard treatment — The treatment to be used in the study is in accordance with the latest guidelines for chronic LBP [George et al., 2021; Owen, et al., 2020]. A warm-up will be performed by walking on a treadmill for 10 minutes, followed by 3 sets of 10 to 15 repetitions of exercise: bridge, cat, abdominal, straight leg raising, and oyster, and 3 sets of 30 to 60 seconds of each isometric exercise (front plank and side plank), where the therapist will assess the optimal amount of repetitions for each individual. The rest period between sets will be 40 seconds, and the rest period between exercises will be 1 minute. The total duration of the session will be 40 minutes [Sipaviciene et al., 2020; Kim et al, 2020].
  Arms: Standard treatment
Other: Osteopathy treatment — The osteopathy treatment group (OTG) will receive the same standard treatment for low back pain as the STG, which will be applied twice a week and osteopathy treatment every 15 days for 8 weeks, totaling 4 sessions. The duration of the osteopathy sessions
  Arms: Osteopathy treatment

SUMMARY:
Background: Low back pain is one of the most common musculoskeletal health problem with the highest prevalence in the adult population; globally, it represents a relevant cause of medical, social and economic burden. The aim of the proposed study is to determine the effect of a standard treatment for non-specific low back (CNSLBP) combined with multimodal osteopathy treatment on pain intensity and functional capacity.

Methods: This will be a blind randomized clinical trial, with 44 patients with CNSLBP, randomly assigned into two groups: Experimental group (EG) treated with therapeutic exercises and multimodal osteopathy treatment (n=22) and Control group (CG) treated with therapeutic exercises (n=22). Participants will receive treatment twice a week (total of 16 sessions). The primary outcome is pain, measured by numeric rating scale (NRS: score 0-11 points). Secondary outcomes are: Patient-specific functional scale (scored from 0 to 30), Oswestry Disability Questionnaire (ODQ), finger-to-floor distance test (FFD). Participants will be evaluated pre- and post-treatment and after 1 and 3 months (follow-up).

Results: Analysis will be by intention to treat using linear mixed models. Comparisons between groups before and after treatment will demonstrate whether osteopathy treatment exerts a supplementary effect on pain and functional capacity in patients with CNSLBP. The data will be published after the study is completed. The study will support the practice of evidence-based physical therapy for individuals with CNSLBP.

ELIGIBILITY:
Inclusion Criteria:

* Individuals within the age range of 18-70 years;
* Chronic low back pain in the region between the 12th rib and the gluteal fold, with a minimum duration of 6 weeks with or without referral of pain in the lower limbs;
* no specific cause detectable, such as infection, neoplasia, metastasis, osteoporosis, rheumatoid arthritis, fracture, inflammatory process or radicular syndrome.
* baseline pain: minimum intensity score of 3 out of 10 (0 = no pain, 10 = most intense pain) considered and verified by the Numerical Pain Rating Scale (NPRS).

Exclusion Criteria:

* Previous history of spinal disorders (local trauma, cauda equina syndrome, spinal canal stenosis, congenital abnormalities tumor);
* Inflammatory or infectious diseases (rheumatoid arthritis, fibromyalgia and vertebral osteomyelitis);
* Previous lumbar spine surgery;
* Pregnant women;
* Regular opioid analgesics (≥2 times per week) or opioid patches;
* Receiving disability benefits for back pain or even for another health reason;
* Previous injections for back pain, such as facet joint blocks, nerve root or epidural steroid injection in the previous year;
* Having undergone physical therapy, massage, acupuncture or any other therapeutic intervention for back pain in the previous two weeks;
* Osteopathy techniques that are not used as a treatment for low back pain;
* Neuropathic pain tested with Laségue and Valsalva clinical tests.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline and one week and 3 months (follow-up).
  Changes in pain intensity, will be assessed using the NPRS (Numerical Pain Rating Scale). This is an 11-point scale where 0 means "no pain" and 10 means "worst possible pain". NPRS outcome measures will be evaluated pre- and post-treatment.

SECONDARY OUTCOMES:
Disability caused by low back pain | Baseline and one week
  Oswestry Disability Questionnaire (ODQ) will be used to measure disability caused by low back pain. The ODQ is a 10-item scale with higher numbers indicating greater disability. The questionnaire is self-report and includes the following groups of questions: pain intensity and its effect on personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and travelling. Each subscale contains 6 questions and to each question a score from zero to four is assigned. The levels of disability are determined according to the total score as: no disability (0 to 4), mild disability (5 to 14), moderate disability (15 to 24), severe disability (25 to 34), and complete disability (35 to 50).
Lumbar mobility | Baseline and one week
  Finger-to-floor distance (FFD) will be used to assess lumbar mobility in flexion.
Patient-Specific Functional Scale | Baseline and one week
  Patients were asked to identify up to three important activities they were having difficulty with or were unable to perform due to their condition (e.g., low back pain). The assessment was conducted using an 11-point scale (ranging from 0 "unable to perform activity" to 10 "able to perform activity at pre-injury level") .
Prognostic Risk Assessment | Baseline and one week
  The risk of poor prognosis among participants with low back pain, influenced by physical and psychosocial factors, was evaluated using the STarT Back Screening Tool (SBST). The SBST is a 9-item questionnaire that stratifies patients with low back pain into three risk groups (low, medium, and high) that represent their prognosis regarding disability

CONTACTS AND LOCATIONS:
Locations (1):
- Nove de Julho University, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George SZ, Fritz JM, Silfies SP, Schneider MJ, Beneciuk JM, Lentz TA, Gilliam JR, Hendren S, Norman KS. Interventions for the Management of Acute and Chronic Low Back Pain: Revision 2021. J Orthop Sports Phys Ther. 2021 Nov;51(11):CPG1-CPG60. doi: 10.2519/jospt.2021.0304. PMID 34719942
- [Background] Kim B, Yim J. Core Stability and Hip Exercises Improve Physical Function and Activity in Patients with Non-Specific Low Back Pain: A Randomized Controlled Trial. Tohoku J Exp Med. 2020 Jul;251(3):193-206. doi: 10.1620/tjem.251.193. PMID 32669487
- [Background] Owen PJ, Miller CT, Mundell NL, Verswijveren SJJM, Tagliaferri SD, Brisby H, Bowe SJ, Belavy DL. Which specific modes of exercise training are most effective for treating low back pain? Network meta-analysis. Br J Sports Med. 2020 Nov;54(21):1279-1287. doi: 10.1136/bjsports-2019-100886. Epub 2019 Oct 30. PMID 31666220
- [Background] Sipaviciene S, Kliziene I. Effect of different exercise programs on non-specific chronic low back pain and disability in people who perform sedentary work. Clin Biomech (Bristol). 2020 Mar;73:17-27. doi: 10.1016/j.clinbiomech.2019.12.028. Epub 2020 Jan 3. PMID 31923778